CLINICAL TRIAL: NCT02361502
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Comparison Clinical Study to Investigate the Efficacy and Safety of the β3 Adrenoceptor Agonist, Mirabegron With Overactive Bladder Symptoms in Men
Brief Title: MIrabegron With oveRACtive bLadder Symptoms in mEn
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Soo Woong Kim, MD, Seoul National University Hospital, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIRACLE
Record Dates: First submitted 2014-12-11; First posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- placebo (Placebo Comparator): mirabegron placebo qd
  Interventions: Drug: placebo
- mirabegron (Experimental): mirabegron 50mg qd
  Interventions: Drug: mirabegron

INTERVENTIONS:
Drug: mirabegron
  Arms: mirabegron
Drug: placebo
  Arms: placebo

SUMMARY:
The proportion of male patients who participated in the phase III study of mirabegron was about 28% and the data on the efficacy and safety of mirabegron in Korean male OAB patients have limits. For this reason, this study will assess the efficacy and safety of mirabegron in Korean male OAB patients.

DETAILED DESCRIPTION:
About 50 to 75% of men with LUTS secondary to BPH also have overactive bladder symptoms. As a major drug for the treatment of overactive bladder symptoms, muscarinic receptor antagonists are used, but precautions should be taken by a specialist when using muscarinic receptor antagonists due to possibilities of dry mouth, constipation, blurred vision and post-dose dysuria and acute ischuria. Mirabegron is a selective β3-adrenoceptor agonist that relax the detrusor smooth muscle and increase functional bladder capacity to improve overactive bladder symptoms. This study will examine the efficacy and safety of mirabegron, a new drug, for improvement of urinary frequency.

The efficacy of mirabegron compared to the placebo has been demonstrated by the phase III study, but the analysis of only patients in Korea has not obtained significant difference from the placebo. The prevalence of overactive bladder was 9.7% in men and 11.6% in women, which showed similar rates 1), but the cure rate is higher in men than in women (OR 1.891, CI 1.362, 2.2627, p=0.0001). Male patients are important customers for the OAB market and low-dose anticholinergic agents with relatively low risk of urinary retention are preferred for the treatment of male overactive bladder (OAB) in Korea. We will conduct this clinical study because we think mirabegron will be an alternative for the therapy for male OAB patients with a risk of urinary retention.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 20 years
* Patients with an average of at least 8 micturitions per 24 hours in last 3 days based on the micturition diary
* Patients with an average of at least 1 episode of urgency per 24 hours in last 3 days based on the micturition diary
* Patients who have symptoms of OAB for at least 12 weeks prior to the enrollment
* Patients who are able to complete the micturition diary and questionnaires correctly
* Patients who provided a singed consent form after being informed of the nature of the study and risk and benefit of the study treatment.

Exclusion Criteria:

* Patients with AUR history
* Patients with PSA ≥ 10 ng/ml or suspected prostate cancer
* Patients who have an average total daily urine volume ≥ 3000 mL
* Patients with suspected stress incontinence
* Patients with PVR ≥200 ml or Qmax ≤5ml/sec
* Patients who have used according to the criteria below:

  * Patients who began or discontinued the drug(s) or changed the dose within 4 weeks before enrollment
  * Patients who were treated with an anticholinergic agent, 5-aplha reductase inhibitor within 4 weeks before enrollment
  * Patients who began or discontinued 5ARI treatment or changed the dose within 6 months
* Patients began or has changed a bladder training program or pelvic floor exercises less than 4 weeks prior to Screening.
* Patients who had an indwelling catheter or practices intermittent self-catheterization
* Patients who received surgical treatment that may influence urinary track function (TURP, laser therapy, etc.) within 24 weeks of run-in period
* Uncontrolled hypertension: SBP ≥180 mmHg, DBP ≥110 mmHg
* Pulse rate ≥110 bmp or <50 bpm
* Patients with complications of urinary tract infection, urolithiasis and interstitial cystitis or past history of recurrent urinary tract infection
* Patients with hypersensitivity to β-adrenergic receptor agonists or anticholinergics
* Patients has a clinically significant ECG abnormality, as determined by the Investigator

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean number of micturitions per 24 hours | after 12 weeks of treatment

SECONDARY OUTCOMES:
Change in mean number of urgency episodes per 24 hours | after 12 weeks of treatment
Change in mean number of urgency incontinence episodes per 24 hours | after 12 weeks of treatment
Change in a total of OABSS | after 12 weeks of treatment
Change in residual volume and maximal urinary flow rate | after 12 weeks of treatment
Change in IPSS storage subscore | after 12 weeks of treatment
Change in IPSS-QOL symptom score | after 12 weeks of treatment
Number of Adverse Events of study drug | after 12 and 24 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (14):
- South Korea (14):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Korea University Ansan Hospital, Ansan
  - Pusan National University Hospital, Busan
  - Kyung kook University Hospital, Daegu
  - Eulji University Hospital, Daejeon
  - Ga-cheon University Gil Hospital, Incheon
  - Cheonnam University Hospital, Kwangju
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Kang book Samsung Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul